CLINICAL TRIAL: NCT02355262
Title: Community-Based HIT Tools for Cancer Screening and Health Insurance Promotion (CATCH-UP)
Brief Title: CATCH-UP Intervention in Increasing Cancer Screening and Prevention Care in Uninsured Patients at Community Health Centers
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Kaiser Permanente (Other); National Cancer Institute (NCI) (NIH); Oregon Community Health Information Network (Unknown); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jennifer Devoe, MD, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: IRB00009862; NCI-2014-02326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CR00024554; 5219; MR00042926; MR00044877; IRB00009862 (Other: OHSU Knight Cancer Institute); R01CA181452 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-02-04 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Breast Carcinoma; Cervical Carcinoma; Colorectal Carcinoma; Health Status Unknown; Human Papillomavirus Infection; Malignant Neoplasm
Keywords: Insurance Coverage; Insurance Continuity
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Papillomavirus Infections; Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Arm I (Independent Tool Implementation): Participants receive CATCH-UP tools which include a panel management/data aggregator system that identifies patients who may be eligible for public coverage but are not yet insured, or who are nearing coverage expiration, coupled with automated patient outreach and communication at baseline.
  Interventions: Other: Informational Intervention
- Arm II (Tool Implementation with Interactive Facilitation): Participants receive CATCH-UP tools which include a panel management/data aggregator system that identifies patients who may be eligible for public coverage but are not yet insured, or who are nearing coverage expiration, coupled with automated patient outreach and communication. Participants also receive additional implementation support such as trainings, assistance with workflows, and practice facilitation.
  Interventions: Other: Informational Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive CATCH-UP intervention

SUMMARY:
This randomized research trial studies the Community-based Health Information Technology (HIT) Tools for Cancer Screening and Health Insurance Promotion (CATCH-UP) intervention in increasing cancer screening and prevention care in uninsured patients at community health centers. The CATCH-UP intervention may contribute to increased rates of insurance coverage, leading to improved cancer screening and prevention rates in community health care settings, and general recommended preventive care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of the CATCH-UP intervention on up-to-date status of cancer screening and preventive care received by patients.

II. Evaluate the effect of the CATCH-UP intervention on patients? insurance coverage rates.

III. Evaluate the intervention implementation process, patient and community health center (CHC) staff acceptance and use of the CATCH-UP tools, and the patient-, provider-, and system-level factors associated with successful implementation and sustainability of the tools, using mixed methods.

OUTLINE: CHC clinics are randomized to 1 of 2 groups. We compare between groups and with a matched-comparison group.

GROUP I (INTERVENTION ARM 1): Participants receive CATCH-UP tools which include a panel management/data aggregator system that identifies patients who may be eligible for public coverage but are not yet insured, or who are nearing coverage expiration, coupled with automated patient outreach and communication at baseline.

GROUP II (INTERVENTION ARM 2): Participants receive CATCH-UP tools which include a panel management/data aggregator system that identifies patients who may be eligible for public coverage but are not yet insured, or who are nearing coverage expiration, coupled with automated patient outreach and communication. Participants also receive additional implementation support such as trainings, assistance with workflows, and practice facilitation.

Matched-comparison group: A clinic-level matched comparison group will be derived from the OCHIN membership by using propensity score matching techniques. Comparison group clinics will not participate actively in any study activities but, as part of their member business associate agreement with OCHIN, have already agreed to provide data through OCHIN for pre- and post-implementation analysis in the study.

ELIGIBILITY:
Inclusion Criteria:

* Established patients at CHC sites
* Low-income
* Ethnically diverse populations with lower rates of cancer screening compared to national rates
* Uninsured patients
* Patients 18 to 64 years of age
* Clinics must be primary care sites, with greater than 1,000 adult patients in the past year, be located in a state that expanded Medicaid, and have implemented the OCHIN EHR prior to January 1, 2012

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with at least one encounter at a CHC in the OCHIN network since January 1, 2012
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in the proportion of clinic patients who receive age- and gender-appropriate recommended cancer screening and preventive care (clinic-level) | Baseline to up to 6 years
  Pre- and post-implementation differences in proportion of patients with insurance continuity will be calculated between implementation and control community health centers (?difference-in-differences? analysis). Generalized linear/non-linear mixed models will be used, which offer flexible regression modeling to accommodate different sources of correlations (serial and intra-clinic), categorical and continuous covariates, and fixed and time-dependent covariates.
Changes in the proportion of clinic patients with insurance continuity | Baseline to up to 6 years
  Pre- and post-implementation differences in proportion of patients with insurance continuity will be calculated between implementation and control community health centers (?difference-in-differences? analysis). Generalized linear/non-linear mixed models will be used, which offer flexible regression modeling to accommodate different sources of correlations (serial and intra-clinic), categorical and continuous covariates, and fixed and time-dependent covariates. Serial and intra-clinic correlations will be modeled as random effects.
Total number of months uninsured (total gap months) | Up to 6 years
  The Community-based Health Information Technology (HIT) Tools for Cancer Screening and Health Insurance Promotion tool?s impact on total number of months uninsured (total gap months) will be evaluated. The distribution of total gap months will be examined before selecting a specific model to use for the analysis. Analytic models will be refined through an iterative process, guided by the hypotheses and preliminary analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DeVoe, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Background] Hoopes MJ, Angier H, Gold R, Bailey SR, Huguet N, Marino M, DeVoe JE. Utilization of Community Health Centers in Medicaid Expansion and Nonexpansion States, 2013-2014. J Ambul Care Manage. 2016 Oct-Dec;39(4):290-8. doi: 10.1097/JAC.0000000000000123. PMID 26765808
- [Background] Hatch B, Tillotson C, Angier H, Marino M, Hoopes M, Huguet N, DeVoe J. Using the electronic health record for assessment of health insurance in community health centers. J Am Med Inform Assoc. 2016 Sep;23(5):984-90. doi: 10.1093/jamia/ocv179. Epub 2016 Jan 23. PMID 26911812
- [Background] DeVoe JE, Tillotson CJ, Marino M, O'Malley J, Angier H, Wallace LS, Gold R. Trends in Type of Health Insurance Coverage for US Children and Their Parents, 1998-2011. Acad Pediatr. 2016 Mar;16(2):192-9. doi: 10.1016/j.acap.2015.06.009. Epub 2015 Aug 18. PMID 26297668
- [Background] DeVoe JE, Huguet N, Likumahuwa-Ackman S, Angier H, Nelson C, Marino M, Cohen D, Sumic A, Hoopes M, Harding RL, Dearing M, Gold R. Testing health information technology tools to facilitate health insurance support: a protocol for an effectiveness-implementation hybrid randomized trial. Implement Sci. 2015 Aug 25;10:123. doi: 10.1186/s13012-015-0311-4. PMID 26652866
- [Background] Angier H, Hoopes M, Gold R, Bailey SR, Cottrell EK, Heintzman J, Marino M, DeVoe JE. An early look at rates of uninsured safety net clinic visits after the Affordable Care Act. Ann Fam Med. 2015 Jan-Feb;13(1):10-6. doi: 10.1370/afm.1741. PMID 25583886
- [Background] Heintzman J, Marino M, Hoopes M, Bailey SR, Gold R, O'Malley J, Angier H, Nelson C, Cottrell E, Devoe J. Supporting health insurance expansion: do electronic health records have valid insurance verification and enrollment data? J Am Med Inform Assoc. 2015 Jul;22(4):909-13. doi: 10.1093/jamia/ocv033. Epub 2015 Apr 17. PMID 25888586
- [Background] DeVoe JE, Angier H, Burdick T, Gold R. Health information technology: an untapped resource to help keep patients insured. Ann Fam Med. 2014 Nov-Dec;12(6):568-72. doi: 10.1370/afm.1721. PMID 25384821
- [Background] Gold R, Burdick T, Angier H, Wallace L, Nelson C, Likumahuwa-Ackman S, Sumic A, DeVoe JE. Improve Synergy Between Health Information Exchange and Electronic Health Records to Increase Rates of Continuously Insured Patients. EGEMS (Wash DC). 2015 Aug 6;3(1):1158. doi: 10.13063/2327-9214.1158. eCollection 2015. PMID 26355818
- [Background] Huguet N, Hoopes MJ, Angier H, Marino M, Holderness H, DeVoe JE. Medicaid Expansion Produces Long-Term Impact on Insurance Coverage Rates in Community Health Centers. J Prim Care Community Health. 2017 Oct;8(4):206-212. doi: 10.1177/2150131917709403. Epub 2017 May 17. PMID 28513249
- [Derived] Huguet N, Valenzuela S, Marino M, Moreno L, Hatch B, Baron A, Cohen DJ, DeVoe JE. Effectiveness of an insurance enrollment support tool on insurance rates and cancer prevention in community health centers: a quasi-experimental study. BMC Health Serv Res. 2021 Oct 30;21(1):1186. doi: 10.1186/s12913-021-07195-5. PMID 34717616
- [Derived] Hatch B, Tillotson C, Huguet N, Marino M, Baron A, Nelson J, Sumic A, Cohen D, E DeVoe J. Implementation and adoption of a health insurance support tool in the electronic health record: a mixed methods analysis within a randomized trial. BMC Health Serv Res. 2020 May 15;20(1):428. doi: 10.1186/s12913-020-05317-z. PMID 32414376